CLINICAL TRIAL: NCT03844763
Title: The CONFRONT Phase I - II Trial: ACtivatiON oF Immune RespONse in paTients With R-M Head and Neck Cancer. Multimodality Immunotherapy With Avelumab, Short Course Radiotherapy and Cyclophosphamide in Head and Neck Cancer.
Brief Title: Targeting the Tumor Microenvironment in R/M SCCHN
Acronym: CONFRONT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-000353-39
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: Immunotherapy; Avelumab; Head and neck cancer; Radiotherapy; Cyclophosphamide
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — avelumab; Cyclophosphamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I - II trial of CTX, RT, Avelumab (Experimental): CTX: 50 mg Daily untill PD or major toxicity; Avelumab: 10 mg/kg every 2 weeks, untill PD or major toxicity; RT: 8 Gy single shot day 8.
  Interventions: Drug: Avelumab; Drug: CTX; Radiation: RT

INTERVENTIONS:
Drug: Avelumab — Avelumab: 10 mg/kg every 2 weeks, untill PD or major toxicity
  Other Names: anti PD-L1
Drug: CTX — CTX: 50 mg Daily untill PD or major toxicity
  Other Names: cyclophosphamide
Radiation: RT — RT: 8 Gy single shot day 8
  Other Names: Radiotherapy

SUMMARY:
Phase I - II trial of the combination of cyclophosphamide, RT, and Avelumab in relapsed/metastatic HNSCC (R/M-HNC). Patients pretreated with at least one line therapy containing platinum, fluorouracil, and Cetuximab. Treatment consists of metronomic cyclophosphamide 50 mg daily without drug free break, avelumab 10 mg/kg d1 and 15 q 29, and radiotherapy in one or three daily fractions up to 8 Gy maximum dose, starting at day 8. The aim of the study is to reverse tumor immune-escape by:

1. Provide a self-vaccination with radiotherapy
2. Inhibit the immunosuppressive CD4+ CD25+ FoxP3+ Treg cells with metronomic cyclophosphamide
3. Reactivate the effector T cell by the inhibition of PD-1 - PD-L1 axis with avelumab.

Due to the supposed biological effects of the present trial, an ancillary translational study is needed and will be extended to all the patients' population enrolled.

DETAILED DESCRIPTION:
Rational of the trial

A phase I - II trial in RM-HNC based on pharmacologic and physic interventions related to each other facing immunology as a system rather than a single pathway, theoretically able to restore immune competence toward the tumor. The immune suppressive mechanisms that could be affected by this study and how the experimental approach could inhibit them, are listed below:

* PD-1 - PD-L1 axis is widespread among immune cell family including CTL, Treg, NK, NKT, APC and others showing, for example, opposite effect in CD8+ CTL (inhibitory signal) or in CD4+ CD25+ Foxp3+ (activating signal).
* Depletion of Treg results in tumor regression, in experimental models. The effect seems to be dependent on the extent of Treg suppression.
* Avelumab is a fully human anti-PD-L1 IgG1 monoclonal antibody. It enables the activation of T-cells and the adaptive immune system by inhibiting PD-1 - PD-L1 axis, induces antibody-dependent cell-mediated cytotoxicity (ADCC) and engages the innate immune system.
* Low dose cyclophosphamide (metronomic cyclophosphamide), selectively reduce Treg population both in experimental models and in humans, but it does not affect effector T cells
* PD-1 - PD-L1 axis enhances and sustains Foxp3 expression and the suppressive function of inducible Tregs (iTrge)7. The blockade of the PD1 - PDL1 axis by Avelumab may have an opposite effect.
* The contemporary use of two, independent, mechanisms of Treg control (Avelumab inhibiting Treg clonal expansion and functions, and cyclophosphamide reducing Treg population) may result in a profound inhibition of Treg population.
* If the suppressive mechanisms of the immune system are weakened, the release of high quantity of tumor specific antigens or stress related antigens (epcam, HSPs, HMBG-1, Calreticulin, ATP), obtained by the induction of immunogenic cell death may induce a sort of "self vaccination" resulting into an effective immune response.
* Radiation may induce immunogenic cell death even in heavily pretreated patients in whom the use of cytotoxic chemotherapy may not, due to the previous exposure to drugs and the development of resistance mechanisms. More precisely, this effect is considered the basis of the Abscopal effect, i.e. the regression of tumor deposits outside the irradiated field. This effect is more frequently observed with low-dose, non ablative, hypofractionated radiation therapy (described at point 2.3.2) and represent a proof of concept that in particular situations, radiotherapy act as an inducer of "self vaccination".
* IgG1 mAbs, such as Avelumab, triggers ADCC; PD-L1 is widely express in many tumors and so ADCC may represent an additional mechanism of tumor control.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial. The subject may also provide consent for the translational study.
2. Be 18 years of age on day of signing informed consent.
3. ECOG Performance Status 0-2.
4. Have histologically or cytologically-confirmed recurrent or metastatic (disseminated) head and neck squamous cell carcinoma
5. Have a disease progression after treatment with at least one line of therapy including at least Cisplatin, Fluorouracil and Cetuximab for recurrent (disease not amenable to curative treatment)/metastatic disease.
6. Measurable disease by RECIST criteria.
7. At least one metastatic site suitable for irradiation
8. Life expectancy > 3 months.
9. Adequate bone marrow function: neutrophils 1.5 x 109/L, platelets 100 x 109/L, hemoglobin 9 g/dL.
10. Adequate liver function: AST and ALT levels 2.5 × ULN; bilirubin 1.5 x ULN.
11. Adequate renal function: creatinine clearance 30 mL/min (Cockroft-Gault).
12. Fertil men must be using adequate contraceptive measures throughout the study period if their partner are women of childbearing potential.
13. If of childbearing potential, women must use effective contraceptive method (Pearl Index < 1; e.g. oral contraceptive (pill), hormone spiral, hormone implant, transdermal patch, a combination of two barrier methods (condom and diaphragm), sterilisation, sexual abstinence) for the study duration and for at least 6 months after last avelumab treatment administration if the risk of conception exists.

Exclusion Criteria:

1. History of malignant disease (with the exception of non-melanoma skin tumours and/or in situ cervical cancer) in the preceding five years.
2. Brain metastases.
3. Autoimmune disorders. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
4. Allergic disorders.
5. Cyclophosphamide treatment contraindications:

   1. Cystitis.
   2. Urinary Obstruction.
   3. Inadequate bone marrow function: WBC <2900 mm3 and/or HCT <30% and/or platelets count <90000 mm3.
   4. Active infections.
   5. Pregnancy or breast feeding.
6. Prior treatment with inhibitors of the PD-L1 - PD - 1 axis or inhibitors of CTLA-4 (immune check point inhibitors)
7. Previous HBV or HCV infections.
8. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. systemic corticosteroids at physiologic doses 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
9. Any active infection requiring specific treatment (Antibiotics, antimicotic, antiviral).
10. Radiotherapy within 6 weeks before enrolment
11. Other non-malignant uncontrolled systemic diseases or social conditions that would preclude trial entry in the opinion of the investigator.
12. Prior organ transplantation including allogenic stem-cell transplantation.
13. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
14. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade 2, or other Grade 2 not constituting a safety risk based on investigator's judgment are acceptable.
15. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
16. Avelumab treatment contraindications:

    1. Hypersensitivity to the active ingredient or to any excipient.
    2. Inadequate bone marrow function: WBC <2900 mm3 and/or HCT <30% and/or platelets count <90000 mm3.
    3. Uncontrolled serous effusions (pleural, pericardic or peritoneal)
    4. Blood Pressure <60 mmHg.
    5. Pregnancy or breast feeding.
    6. Active infections. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
    7. Brain metastases.
    8. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure ( New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
17. Participation to other concomitant experimental study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 4 months
  Assessment of the safety profile of the association of avelumab and metronomic cyclophosphamide will be graded using the common toxicity criteria and adverse events (NCI CTC-AE v 4.0).Grade refers to the severity of the AE. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. Each adverse event will be reported as the maximum level observed in each patient.
Objective response rate | 2-4 months
  Objective response is defined as complete response or partial response as defined as per RECIST evaluation criteria v1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Toxicity of the combination | 1 month
  Assessment of the safety profile of the association of avelumab and metronomic cyclophosphamide will be graded using the common toxicity criteria and adverse events (NCI CTC-AE v 4.0).Grade refers to the severity of the AE. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE. Each adverse event will be reported as the maximum level observed in each patient.
Progression Free Survival (PFS) | 54 months
  Progression free survival is defined as the time from study treatment initiation to the first occurrence of disease progression or death of any cause, whichever occurs first.
Quality of Life (QoL) | 2 months
  Quality of Life will be assessed using the EORTC QLQ -30. Grade 1 to 4. Grade 1: not at all, Grade 4: Very much
H&N specific Quality of Life (QoL) | 2 months
  Quality of Life will be assessed using the EORTC QLQ - H&N35. Grade 1 to 4. Grade 1: not at all, Grade 4: Very much
Overall Survival (OS) | 54 months
  Overall survival is defined as the time from treatment initiation to death for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: MARCO C MERLANO, DR, Principal Investigator — AO S CROCE E CARLE DI CUNEO
Locations (2):
- Italy (2):
  - AO Santa Croce e Carle di Cuneo, Cuneo, Italia/cuneo
  - Azienda Ospedaliera S. Croce E Carle Di Cuneo - Cuneo (Cn) Oncologia Medica, Cuneo

REFERENCES:
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Intlekofer AM, Thompson CB. At the bench: preclinical rationale for CTLA-4 and PD-1 blockade as cancer immunotherapy. J Leukoc Biol. 2013 Jul;94(1):25-39. doi: 10.1189/jlb.1212621. Epub 2013 Apr 26. PMID 23625198
- [Background] Francisco LM, Salinas VH, Brown KE, Vanguri VK, Freeman GJ, Kuchroo VK, Sharpe AH. PD-L1 regulates the development, maintenance, and function of induced regulatory T cells. J Exp Med. 2009 Dec 21;206(13):3015-29. doi: 10.1084/jem.20090847. Epub 2009 Dec 14. PMID 20008522
- [Background] Li X, Kostareli E, Suffner J, Garbi N, Hammerling GJ. Efficient Treg depletion induces T-cell infiltration and rejection of large tumors. Eur J Immunol. 2010 Dec;40(12):3325-35. doi: 10.1002/eji.201041093. PMID 21072887
- [Background] Ghiringhelli F, Menard C, Puig PE, Ladoire S, Roux S, Martin F, Solary E, Le Cesne A, Zitvogel L, Chauffert B. Metronomic cyclophosphamide regimen selectively depletes CD4+CD25+ regulatory T cells and restores T and NK effector functions in end stage cancer patients. Cancer Immunol Immunother. 2007 May;56(5):641-8. doi: 10.1007/s00262-006-0225-8. Epub 2006 Sep 8. PMID 16960692
- [Background] Haikerwal SJ, Hagekyriakou J, MacManus M, Martin OA, Haynes NM. Building immunity to cancer with radiation therapy. Cancer Lett. 2015 Nov 28;368(2):198-208. doi: 10.1016/j.canlet.2015.01.009. Epub 2015 Jan 12. PMID 25592036
- [Background] Chandra RA, Wilhite TJ, Balboni TA, Alexander BM, Spektor A, Ott PA, Ng AK, Hodi FS, Schoenfeld JD. A systematic evaluation of abscopal responses following radiotherapy in patients with metastatic melanoma treated with ipilimumab. Oncoimmunology. 2015 May 28;4(11):e1046028. doi: 10.1080/2162402X.2015.1046028. eCollection 2015 Nov. PMID 26451318

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT03844763/Prot_SAP_000.pdf